CLINICAL TRIAL: NCT06970951
Title: A Single-Arm, Open-Label, Single-Center Investigator-Initiated Early-Stage Clinical Study for Relapsed/Refractory (R/R) Autoimmune Diseases
Brief Title: Early Clinical Study of UTAA91 Injection for the Treatment of Relapsed/Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-009-03
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis; Dry Syndrome; Idiopathic Inflammatory Myopathies; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Myositis; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: UTAA91 injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTAA91 injection (Experimental): Infusion of UTAA91 injection in subjects screened after signing informed consent.
  Interventions: Biological: UTAA91 injection

INTERVENTIONS:
Biological: UTAA91 injection — Infusion of UTAA91 injection in subjects screened after signing informed consent.

SUMMARY:
This clinical trial is designed as a single - arm, open - label, single - center, investigator - initiated early - phase clinical study. The primary objective is to evaluate the safety of UTAA91 injection in treating subjects with relapsed/refractory autoimmune inflammatory diseases (AID).

DETAILED DESCRIPTION:
Following the signing of the informed consent form, eligible subjects will receive an infusion of UTAA91 injection. Blood samples will be collected from the subjects before and after the infusion for pharmacokinetic, pharmacodynamic, immunogenicity, and safety assessments.

Aside from the baseline period, efficacy evaluations will be conducted periodically during the treatment phase after cell reinfusion until the occurrence of one of the following events, with the earliest event taking precedence: disease progression, initiation of new anti - disease treatment, death, intolerable toxicity, the investigator's decision, or the subject's voluntary withdrawal.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years (including the cut - off value), with no restrictions on gender.
2. Expected survival time ≥ 3 months.
3. Subjects with relapsed/refractory autoimmune diseases who have failed standard treatment or lack effective treatment options, including but not limited to rheumatoid arthritis, systemic sclerosis, systemic lupus erythematosus, idiopathic inflammatory myopathies, Sjögren's syndrome, connective tissue disease - related interstitial lung disease, immune thrombocytopenia, primary biliary cholangitis, etc.
4. Liver and kidney functions and cardiopulmonary functions meet the requirements.
5. No severe mental disorders.
6. Able to understand this trial and have signed the informed consent form.

Exclusion Criteria

1. Malignant tumors other than relapsed/refractory autoimmune diseases (R/R AID) within 5 years before screening.
2. Subjects with positive virus and/or syphilis tests.
3. Presence of severe heart disease or unstable systemic diseases.

5. Presence of active or uncontrollable infections requiring systemic treatment.

6. Pregnant or breastfeeding women, as well as female subjects who plan to become pregnant within 2 years after cell infusion or male subjects whose partners plan to become pregnant within 2 years after their cell infusion.

7. Subjects who have received CAR - T therapy or other gene - modified cell therapies before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | About 1 year
  The types, frequency, and severity of adverse events (AEs) and laboratory abnormalities (according to the Common Terminology Criteria for Adverse Events, NCI CTCAE 5.0).

SECONDARY OUTCOMES:
Cmax | About 1 year
  Maximum concentration of UTAA91 injection amplified in peripheral blood after administration of the drug
Tmax | About 1 year
  Time to reach maximum concentration in peripheral blood after administration of UTAA91 injection
Disease remission rate | About 3 months
  The disease remission/response/improvement rates at 28 days, 2 months, and 3 months after treatment with UTAA09 injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wu, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No